CLINICAL TRIAL: NCT01351922
Title: A Cross-Sectional Survey to Evaluate Diabetes Management, Control, Complications, Psychosocial Aspects of Diabetic Patients in India and to Evaluate Perceptions and Practices of Physicians and Patients About Diabetes Management in India (DiabCare India 2011)
Brief Title: A Survey to Evaluate Diabetes Management, Control, Chronic Complications, Psychosocial Aspects of Diabetic Subjects in India
Acronym: DiabCare India
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-3933; U1111-1120-5710 (Other: WHO)
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Patients will fill out a questionaire by interview.

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to evaluate the current status of diabetes management, control, and complications in diabetic subjects in India. Perceptions and practices of physicians and subjects about diabetes management will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have visited the centre at least once in the last 3-6 months apart from the initial visit
* First twenty patients of diabetes visiting the centre during the data collection period
* Patients willing to sign the informed consent form

Exclusion Criteria:

* Repetition of any patient as patients should not be included twice for any reason
* Unwilling to participate or unable to comply with protocol requirements

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diabetes mellitus (both type 1 and type 2) being treated at general hospitals, diabetes clinics and referral clinics will be selected according to inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Mean age of onset of type 1 diabetes mellitus | Evaluation visit
Mean age of onset of type 2 diabetes mellitus | Evaluation visit
Mean duration of treatment of type 2 diabetes mellitus | Evaluation visit
Percentage of patients on Insulin therapy | Evaluation visit
Percentage of patients on Oral Anti-Diabetics Drug (OADs) therapy | Evaluation visit
Mean duration of diabetes in type 1 patients | Evaluation visit
Mean duration of diabetes in type 2 patients | Evaluation visit
Mean FPG (fasting plasma glucose) | Evaluation visit
PPG (post prandial glucose) | Evaluation visit
HbA1c (Glycosylated Haemoglobin) | Evaluation visit
Percentage of patients archiving HbA1c target below or equal 6.5% | Evaluation visit
Percentage of patients archiving HbA1c target below or equal 7.0% | Evaluation visit
Percentage of patients having complications (dyslipidemia and hypertension, cardiovascular complications, peripheral vascular disease, diabetic nephropathy and diabetic eye complications) | Evaluation visit

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bangalore, India

REFERENCES:
- [Result] Mohan V, Shah SN, Joshi SR, Seshiah V, Sahay BK, Banerjee S, Wangnoo SK, Kumar A, Kalra S, Unnikrishnan AG, Sharma SK, Rao PV, Akhtar S, Shetty RV, Das AK; DiabCare India 2011 Study Group. Current status of management, control, complications and psychosocial aspects of patients with diabetes in India: Results from the DiabCare India 2011 Study. Indian J Endocrinol Metab. 2014 May;18(3):370-8. doi: 10.4103/2230-8210.129715. PMID 24944934
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com